CLINICAL TRIAL: NCT05579301
Title: Biomarker Development for Progressive Supranuclear Palsy Through Multi-dimensional SNU-PSP Cohort Database
Brief Title: Study of Comprehensive ANd Multimodal Marker-based Cohort of Progressive Supranuclear Palsy(PSP)
Acronym: SCAN-PSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jee-Young Lee, Clinical Professor, Seoul National University Hospital
Other Study IDs: SNUH_2022_0117
Record Dates: First submitted 2022-06-20; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — For participants enrolled in the cohort, a baseline blood sample will be collected and stored for analyses in the future. Blood will also be stored for high throughput 'omics (transcriptomics, genomics and proteomics) to develop new biomarkers for diagnosis and disease progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSP patients: Patients with PSP according to the inclusion and exclusion criteria
- healthy controls: age-matched healthy controls according to the inclusion and exclusion criteria

SUMMARY:
The purpose of this cohort study is to develop a reliable biomarker in progressive nuclear palsy (PSP).

DETAILED DESCRIPTION:
Progressive supranuclear palsy is a rapidly progressive neurodegenerative disease without a cure. Thus, the development of a biomarker that reflects and monitors disease severity in PSP is critical for early diagnosis and performing a successful clinical trial. Thus, we will prospectively recruit patients with PSP and collect comprehensive clinical, imaging and blood biomarkers at baseline with longitudinal follow-up for 1 year.

ELIGIBILITY:
Inclusion Criteria for the patient group:

* Age 50 to 80 years, male or female
* Progressive supranuclear palsy (PSP) patients who are diagnosed as Probable, Possible or suggestive PSP with Movement Disorder society diagnostic criteria for PSP (Hoglinger et al., 2017)

Exclusion Criteria for the patient group:

* Subjects with clinically significant psychiatric illness
* Subjects with cancer or severe medical illness
* Lactating, pregnant, or possibly pregnant
* Subjects with small vessel disease (> grade II) in brain MRI or other structural lesions by causes other than PSP
* Subjects with severe dementia patients (MMSE < 19 or MoCA <13 or General deterioration scale >= 5)

Inclusion Criteria for the healthy control group:

* Age 50 to 80 years, male or female
* Those who agreed to participate in this study

Exclusion Criteria for the healthy control group:

* Those with a history of any neurological diseases
* Lactating, pregnant, or possibly pregnant
* Subjects with clinically significant psychiatric illness
* Subjects with cancer or severe medical illness

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of Target population
  Patient group: 100, Healthy control group: 30
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-12-19 (Actual); Primary Completion 2024-12-19 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in the Progressive Supranuclear Palsy Rating Scale (PSP-RS) | From the baseline to 6 months and 12 months follow-up
  A scale for assessment of motor and non-motor symptom severity in PSP patients. The PSPRS comprises 28-items with total score ranges from 0 (normal) to 100.

SECONDARY OUTCOMES:
Change in the Schwab & England Activity of Daily Living scale (SEADL) | From the baseline to 6 months and 12 months follow-up
  A scale for activity of daily living assessment that ranges from 0% (complete dependence) to 100% (total independence). The decline in the ADL percentage over time indicates worsening.
Change in cognitive battery for seoul neuropsychological screening battery (SNSB-2) scale | From the baseline to 6 months and 12 months follow-up
  SNSB-2 measures 5 cognitive domain including memory, frontal executive function, attention, visuospatial, language. SNSB scores are provided as age, sex normalized score (z-score) which have a mean of 0 with standard deviation of 1. Higher score indicates better performance.
Change in MoCA (Montreal cognitive assessment) | From the baseline to 6 months and 12 months follow-up
  MoCA scale measures global cognitive status including attention and concentration, executive function, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. MoCA score ranges from 0 to 30. Higher score indicates better performance
Change in MMSE(Mini-mental state examination) | From the baseline to 6 months and 12 months follow-up
  MMSE scale measures global cognitive status that ranges from 0 to 30. Higher score indicates better performance

OTHER OUTCOMES:
FDG PET (18Fluorodeoxyglucose) | From the baseline to 12 months follow-up
  Evaluation of metabolic activity and patterns of the brain
Tau PET (18F-taucipir) | From the baseline to 12 months follow-up
  Evaluation of the tau aggregation in the brain
Structural analysis by 3T MRI | From the baseline to 12 months follow-up
  Evaluation of the degenerative change in the brain
Change in p-tau 181 | From the baseline to 12 months follow-up
  Change in serum and/or plasma phosphorylated tau (p-tau181) in PSP patients
total tau (T-tau) | From the baseline to 12 months follow-up
  Change in serum and/or plasma total tau (T-tau) in PSP patients
Amyloid beta 42 (Aβ-42) | From the baseline to 12 months follow-up
  Change in serum and/or plasma Amyloid beta 42 (Aβ-42) in PSP patients
Proteomic markers | From the baseline to 12 months follow-up
  Change in blood-based proteomic markers
Genomic markers | Baseline
  Identification of genetic markers in PSP that differentiates individuals with different clinical presentation and progression.
Retina biomarkers by OCT imaging | From the baseline to 12 months follow-up
  Exploratory analysis of OCT and OCTA imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jee-Young Lee, M.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (2):
- South Korea (2):
  - Seoul National University Boramae Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No